CLINICAL TRIAL: NCT04432194
Title: Evaluation of the Effect of Nutritional Supplementation and Pulmonary Rehabilitation on the Clinical Status of Patients With Heart Failure and Chronic Obstructive Pulmonary Disease
Brief Title: Effect of Nutritional Supplementation and Pulmonary Rehabilitation on the Clinical Status of HF and COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Dulce González Islas, PhD, Researcher in Medical Sciences, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: C68-18
Record Dates: First submitted 2020-05-25; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure; Copd; Nutritional Supplementation; Pulmonary Rehabilitation
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): The subjects in this group will receive the usual care, which includes the non-pharmacology recommendations by the European Society of Cardiologists 2006 (1) and COPD guides for treatment (6), both founded in the sodium and liquids restriction.
- Pulmonary Rehabilitation Group (Active Comparator): Patients in this group will receive pulmonary rehabilitation specified by rehabilitation doctors according to the needs and capacities of each individual, who will attend three times a week for three months.
  Interventions: Dietary Supplement: Nutritional supplementation and Pulmonary Rehabilitation
- Pulmonary Rehabilitation Group plus HMB (4g) (Experimental): Patients in this group will receive pulmonary rehabilitation specified by rehabilitation doctors according to the needs and capacities of each individual, who will attend three times a week for three months. Furthermore, they will receive 4g of citrulline supplementation.
  Interventions: Dietary Supplement: Nutritional supplementation and Pulmonary Rehabilitation
- Pulmonary Rehabilitation Group plus citrulline (3g) (Experimental): Patients in this group will receive pulmonary rehabilitation specified by the doctor specialized in rehabilitation according to the needs and capacities of each individual, who will attend three times a week for three months. Furthermore, they will receive 4g of citrulline supplementation.
  Interventions: Dietary Supplement: Nutritional supplementation and Pulmonary Rehabilitation

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation and Pulmonary Rehabilitation — Nutritional supplementation (HMB 4g) or Nutritional supplementation (citrulline 3g) with Pulmonary Rehabilitation
  Arms: Pulmonary Rehabilitation Group; Pulmonary Rehabilitation Group plus HMB (4g); Pulmonary Rehabilitation Group plus citrulline (3g)

SUMMARY:
Cardiovascular diseases (CVD) are the leading cause of death in the world and our country. The prevalence of Heart Failure (HF) is 1-2% in the adult population in developed countries, up to 10% among people 70 years of age. Concerning COPD, it is estimated that by 2030 will be the third leading cause of death in the world; the prevalence in Mexico is 18.4%. Also, according to INEGI data, it is the 5th cause of death in people over 65.

50% of patients with COPD die of cardiovascular causes, and they are at higher risk of developing HF, hospital readmissions, and death.

Subjects with HF and COPD concomitant have alterations such as; systemic inflammation, loss of muscle mass and strength of both skeletal and respiratory muscles, reduced tolerance to exercise, and lung function, which has an important impact on clinical status, quality of life and prognosis.

The objective of nutritional treatment in HF is to reduce heart overload and reduce cardiovascular risk. On the other hand, in COPD, it is to improve lung function. However, this is not enough to maintain the protein reserves of patients due to previously affected factors. Therefore, it is vitally essential to contemplate the supplementation with amino acids that prevent and delay the loss of protein reserves, as well as the delay in clinical status.

The β-hydroxy-β-methyl butyrate (HMB) is a metabolite of leucine, with an anticatabolic and anabolic effect. HMB improves the synthesis of proteins, muscle mass, strength, and muscle functionality. Citrulline has been associated with increased muscle mass, VO2, and exercise tolerance.

On the other hand, pulmonary rehabilitation (RP) has improved exercise tolerance, mass, and strength of skeletal and respiratory muscles, quality of life, reduction of hospitalizations, and mortality. However, in concomitant HF and COPD, there are no guidelines that specify the type of RP or if there is a synergistic effect with nutritional supplementation and its impact on clinical status.

DETAILED DESCRIPTION:
Heart Failure

Heart Failure (HF) is a complex syndrome consequence of any structural or functional abnormality that impairs the capacity of filling or ejected of the heart. (1, 2).

Chronic obstructive pulmonary disease

Chronic obstructive pulmonary disease (COPD) is a progressive, systemic, and multi-organic disease with structural and functional changes, mostly in the lungs. It is characterized by a progressive limitation of airflow as a response to external factors such as airflow contamination, smoking, biomass, which are associated with chronic inflammation. (3).

Epidemiology

The cardiovascular disease is the leading cause of death worldwide (4); The HF prevalence goes from 1-2% in developed countries and increases to 10% in older >70 years old.

COPD is an important global load affecting more than 600 million people corresponding to the 5 % off all cause of death worldwide (5).

Chronic Obstructive Pulmonary Disease and Heart Failure

COPD and HF are related between them, sharing the same risk factors and pathogenic mechanisms. They are growing in time and are epidemic diseases because of multiple factors. The cardiovascular disease takes an essential role in COPD, 30 to 50% of deaths are because of them; one of the most important is HF. COPD patients have three times the risk to developed HF (6), and between them, the risk of hospital readmission and death is higher than those without HF (7).

Nutritional Supplementation

β-Hydroxy-β-Methylbutyrate (HMB) HMB is a leucine metabolite, are a branch chain amino acid, and a regular potent in the muscular protein replacement and endogen sub-production that occurs in the muscles and liver. The first stage of change is through the transamination of the leucine to KIC, occurring in the mitochondrial and cytosol of the muscular cell. In the mitochondria, the KIC oxidates into isovaril-CoA, subsequently by other metabolism processes, it produces 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA). Approximately 90% of KIC oxidize into isovaril CoA in the hepatic mitochondrial, lastly, acetoacetate and Acetyl-CoA. While the last 10% oxides into HMB in the cellular cytosol (8-10).

Supplementation with HMB

HMB develops a nutritional role; the daily supplementation has an anti-catabolic effect in the protein synthesis, increasing the muscular mass and diminished the muscular damage in adulthood.

Several studies evaluate the effects of supplementation with HMB, isolated, or combined in muscle functionality, strength, mortality, and indifferent pathologies(11). Recently, in a meth analysis and systemic review of randomized clinical trials made by Wu et al. to evaluate the effect of the administration with HMB over the corporal composition and muscular strength in adulthood in 65 years with pathologies. The study includes supplementation of HMB at 3mg doses at least eight weeks to increase the muscular strength and functionality (12). Supplementation with Ca-HMB with or without resistance exercise in older than 75 years' old was evaluated by Stout et al., in a pilot study, they made 2 phases: the first one (without exercise) supplementation with 3g of CaHMB vs. placebo and the second (with resistance exercise) with and without supplementation. They observed that the supplementation in the long term has better benefits, and increase lean mass, strength, quality, and functional muscle without exercise. In this study, they showed that there is no synergic effect with the exercise combined with supplementation (10).

Citrulline-arginine The principal precursor of citrulline is glutamine, representing 60% of the total synthesis of arginine de novo (13). Citrulline is released into the portal circulation because the enterocytes do not have the succinate arginine synthase. The liver absorbs one quantity in a normal hepatic function and goes to the systemic circulation and finally is transformed by the kidney into arginine (14). The supplementation is a potent nutrient-drug that helps to restore the arginine metabolism in different populations (14, 15).

Citrulline is considered a safe supplementation (16)with a maximum consumption of 15g/day and 13 g/day for arginine (17, 18). The blood levels in a healthy individual are 40 µmol/L (19). L citrulline increases the concentration of L arginine more efficiently than the supplementation of L-arginine; this is an amino acid, endogen precursor of the synthesis of oxide nitric (ON) (20).

Different studies with supplementation show a reduction in adhesion cells and leucocyte activation, as well as an improvement in endothelial function (21). Besides, in heathier subjects, it has been associated with less muscular fatigue, better VO2, and exercise tolerance. (22) In a randomized clinical trial (RCT) with healthy subjects, where they receive oral supplementation with citrulline, they showed an increase of 57% of the nitrogen balance 12 hrs. after (17)

Pulmonary rehabilitation

Pulmonary rehabilitation and physic therapy are essential components of the non-pharmacologic treatment, for HF and COPD, the guidelines' treatment recommends the pulmonary rehabilitation or physic therapy, to improve the exercise tolerance, skeletal and respiratory muscular function, also the quality of life of the patients (23, 24). On the other side, it has been demonstrated that pulmonary rehabilitation and physic therapy have benefits in the number of hospitalization and mortality of patients.

Ancanfora et al., in a randomized clinical trial evaluate the effect of cardiovascular training in patients with HF. The program consists of resistance activities and abdominal exercises, depending on the clinical characteristics of each patient, they were followed by four weeks, resulting in an improvement over-exercise tolerance, O2 maximum consumes and ventilatory threshold (25). Similarly, Keteyian et al., evaluated the physiological adaptation resulting by the physical training in patients with HF with Left ventricle ejection fraction. Also reduced the effects and security in clinical results, had a followed of 2-5 weeks, it consists by resistance exercises such as walking and the use of the static bicycle by 20-30 minutes (23). They conclude that the exercise was secure and improves the state of health, exercise capacity. O´connor et al., evaluated the effects of a regular aerobic exercise (bicycle, treadmill) in patients with HF plus the habitual care, followed by 30 months, they observed that the mortality and hospitalization decreases (26).

Additionally, Benefits have also been seen in patients with COPD; Petersen et al., after seven weeks, show that the resistance exercises twice a week improved exercise tolerance and diminished the fast degradation of proteins (27). Nevertheless, patients with HF and COPD have no guidelines that specified the type of exercise as well as the duration of it, or if there is a synergic effect with nutritional supplementation and which is the impact over the clinic stage.

General objective:

To assess the effect of nutritional supplementation and pulmonary rehabilitation on the clinical status of patients with HF and COPD compared to those subjects who do not receive nutritional supplementation or pulmonary rehabilitation.

Specific objectives

To evaluate the effect of pulmonary rehabilitation and supplementation over body composition in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

To evaluate the effect of pulmonary rehabilitation and supplementation over the exercise tolerance in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

To evaluate the effect of pulmonary rehabilitation and supplementation over pulmonary function in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

To evaluate the effect of pulmonary rehabilitation and supplementation over endothelial function in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

To evaluate the effect of pulmonary rehabilitation and supplementation over muscle function in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

To evaluate the effect of pulmonary rehabilitation and supplementation over cognitive function in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

Evaluated the effect of nutritional supplementation and pulmonary rehabilitation over prognosis in COPD and HF patients compared to those subjects who receive non-pharmacology treatment based on guidelines treatment.

Hypothesis Subjects with HF and COPD who receive nutritional supplementation and pulmonary rehabilitation will have a better clinical status than those who do not receive nutritional supplementation or pulmonary rehabilitation.

Methodology

Design Study:

Randomized clinical trial

Study Population:

Patients with Heart failure and Chronic Obstructive Pulmonary Disease diagnosisStatistical Analysis

Descriptive analysis will be present as frequency and percentage if categorical variables and mean & standard deviation if the variable is continuous with normal distribution; if not, it will report as median and percentiles (25-75). The normality distribution will be evaluated through a Shapiro-Wilk test.

At the beginning of the study, we will compare both groups to determine statistical significance differences. X2 will run in categorical variables and an independent t-study test in continuous variables with normal distribution, if not, U de Mann Whitney will be run.

To identifying the differences between groups along with the study, repeated analysis of variance measures will be done if the variable has a normal distribution. Otherwise, Friedman tests will be made. McNemar will be made for categorical variables. Furthermore, changes between groups along the time at student will be made with a normal distribution; otherwise, Wilcoxon will be done.

Alpha type error: it considered as a statistical significance a p<0.05

Sample size A simple size space of 100 patients, 25 subjects per group will be included if prior consent is acquired, and they meet the inclusion criteria.

Procedures Invitation to participate All the patients who complete the inclusion criteria will be invited to the protocol. They shall be informed about the study, the possible risks and benefits of the treatment, and the possibility of leaving the study at any moment if the patients want. Those who accept participated will be enrolled in a list and then randomized into different groups of treatment.

Allocation to the treatment groups The allocation sequence will be generated in the site http://www.randomization.com; therefore, the patients will be assigned into one of the next groups: 1) control group 2)pulmonary rehabilitation 3) rehabilitation pulmonary group plus beta-hydroxy beta-methyl butyric (HMB) (4g) 4) pulmonary rehabilitation group plus Citrulline (4g). The cardiologist, nutritionist, the physic therapist, will be blinded to the assignation group treatments.

Baseline evaluation During the first evaluation, the clinical stage will be assigned, and the next valuations will be made: pulmonary function, endothelial function, exercise tolerance, functional class, signs, and symptoms. anthropometric and body composition indicators by electric bio-impedance, biochemical test, dietetics, handgrip strength Following visits All the patients, no matter the group, will have a follow up for three months. In the beginning, 6week later and finally at three months.

Survival follow-up wil be after two years treatment initiation

ELIGIBILITY:
Inclusion Criteria:

* Patients that accept and signed the study consent.
* > 40 years old
* Patients with Heart failure diagnosis confirmed by echocardiographic criteria according to the European Society of Cardiology guidelines (2).
* Heart failure patients in functional class I to III according to NYHA
* Patients with Chronic Obstructive Pulmonary Disease diagnosis according to GOLD guidelines with a post-bronchodilator spirometry VEF1/FVC index <0.70 (50)

Exclusion Criteria:

* Patients with recent (<3 months) exacerbations
* Terminal Chronic Renal Kidney Disease with a creatinine clearance <30 ml/min/1.73m2
* Patients with a cancer diagnosis
* Patients with limitation to exercise
* Patients enrolled in another study protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of nutritional supplementation and pulmonary rehabilitation on the clinical status | Baseline, 6 weeks after treatment initiation, 12 weeks 6 weeks after treatment initiation
  Change from baseline in functional class assessed by NYHA
Evaluated the effect of nutritional supplementation and pulmonary rehabilitation over the skeletal muscle mass | Baseline, 6 weeks after treatment initiation, 12 weeks 6 weeks after treatment initiation
  Change from baseline in the skeletal muscle mass assessed by bioelectrical impedance
Evaluated the effect of nutritional supplementation and pulmonary rehabilitation over pulmonary function | Baseline, 6 weeks after treatment initiation, 12 weeks 6 weeks after treatment initiation
  Change from baseline in pulmonary function assessed by spirometry test
To evaluate the effect of pulmonary rehabilitation and supplementation over muscle function in COPD and HF patients | Baseline, 6 weeks after treatment initiation, 12 weeks 6 weeks after treatment initiation
  Change from baseline in pulmonary function assessed by dinamometry test
Evaluated the effect of nutritional supplementation and pulmonary rehabilitation over prognosis in COPD and HF patients | Two years after treatment initiation
  survival follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Verdeja-Vendrell, M.Sc., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas"; Dulce González-Islas, PhD, Study Director — Instituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas"; Arturo Orea-Tejeda, MD, Study Director — Instituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas"; Martha E Quintero-Martínez, B.Sc, Study Chair — Instituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas"; Ilse C Pérez-García, B.Sc, Study Chair — Instituto Nacional de Enfermedades Respiratorias "Ismael Cosío Villegas"
Locations (1):
- Dulce González-Islas, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW. 2009 focused update incorporated into the ACC/AHA 2005 Guidelines for the Diagnosis and Management of Heart Failure in Adults: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the International Society for Heart and Lung Transplantation. Circulation. 2009 Apr 14;119(14):e391-479. doi: 10.1161/CIRCULATIONAHA.109.192065. Epub 2009 Mar 26. No abstract available. PMID 19324966
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. 2016 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure. Rev Esp Cardiol (Engl Ed). 2016 Dec;69(12):1167. doi: 10.1016/j.rec.2016.11.005. No abstract available. English, Spanish. PMID 27894487
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Berger JS, Sanborn TA, Sherman W, Brown DL. Effect of chronic obstructive pulmonary disease on survival of patients with coronary heart disease having percutaneous coronary intervention. Am J Cardiol. 2004 Sep 1;94(5):649-51. doi: 10.1016/j.amjcard.2004.05.034. PMID 15342301
- [Background] Rodriguez LA, Wallander MA, Martin-Merino E, Johansson S. Heart failure, myocardial infarction, lung cancer and death in COPD patients: a UK primary care study. Respir Med. 2010 Nov;104(11):1691-9. doi: 10.1016/j.rmed.2010.04.018. Epub 2010 May 18. PMID 20483577
- [Background] Boudestein LC, Rutten FH, Cramer MJ, Lammers JW, Hoes AW. The impact of concurrent heart failure on prognosis in patients with chronic obstructive pulmonary disease. Eur J Heart Fail. 2009 Dec;11(12):1182-8. doi: 10.1093/eurjhf/hfp148. Epub 2009 Nov 3. PMID 19887495
- [Background] Nissen S, Sharp RL, Panton L, Vukovich M, Trappe S, Fuller JC Jr. beta-hydroxy-beta-methylbutyrate (HMB) supplementation in humans is safe and may decrease cardiovascular risk factors. J Nutr. 2000 Aug;130(8):1937-45. doi: 10.1093/jn/130.8.1937. PMID 10917905
- [Background] Vukovich MD, Stubbs NB, Bohlken RM. Body composition in 70-year-old adults responds to dietary beta-hydroxy-beta-methylbutyrate similarly to that of young adults. J Nutr. 2001 Jul;131(7):2049-52. doi: 10.1093/jn/131.7.2049. PMID 11435528
- [Background] Stout JR, Smith-Ryan AE, Fukuda DH, Kendall KL, Moon JR, Hoffman JR, Wilson JM, Oliver JS, Mustad VA. Effect of calcium beta-hydroxy-beta-methylbutyrate (CaHMB) with and without resistance training in men and women 65+yrs: a randomized, double-blind pilot trial. Exp Gerontol. 2013 Nov;48(11):1303-10. doi: 10.1016/j.exger.2013.08.007. Epub 2013 Aug 24. PMID 23981904
- [Background] Fitschen PJ, Biruete A, Jeong J, Wilund KR. Efficacy of beta-hydroxy-beta-methylbutyrate supplementation in maintenance hemodialysis patients. Hemodial Int. 2017 Jan;21(1):107-116. doi: 10.1111/hdi.12440. Epub 2016 Jun 14. PMID 27302563
- [Background] Rahman A, Wilund K, Fitschen PJ, Jeejeebhoy K, Agarwala R, Drover JW, Mourtzakis M. Elderly persons with ICU-acquired weakness: the potential role for beta-hydroxy-beta-methylbutyrate (HMB) supplementation? JPEN J Parenter Enteral Nutr. 2014 Jul;38(5):567-75. doi: 10.1177/0148607113502545. Epub 2013 Sep 26. PMID 24072740
- [Background] Bahri S, Zerrouk N, Aussel C, Moinard C, Crenn P, Curis E, Chaumeil JC, Cynober L, Sfar S. Citrulline: from metabolism to therapeutic use. Nutrition. 2013 Mar;29(3):479-84. doi: 10.1016/j.nut.2012.07.002. Epub 2012 Sep 28. PMID 23022123
- [Background] Luiking YC, Poeze M, Ramsay G, Deutz NE. Reduced citrulline production in sepsis is related to diminished de novo arginine and nitric oxide production. Am J Clin Nutr. 2009 Jan;89(1):142-52. doi: 10.3945/ajcn.2007.25765. Epub 2008 Dec 3. PMID 19056593
- [Background] Cynober L. Citrulline: just a biomarker or a conditionally essential amino acid and a pharmaconutrient in critically ill patients? Crit Care. 2013 Mar 11;17(2):122. doi: 10.1186/cc12534. PMID 23509945
- [Background] Rouge C, Des Robert C, Robins A, Le Bacquer O, Volteau C, De La Cochetiere MF, Darmaun D. Manipulation of citrulline availability in humans. Am J Physiol Gastrointest Liver Physiol. 2007 Nov;293(5):G1061-7. doi: 10.1152/ajpgi.00289.2007. Epub 2007 Sep 27. PMID 17901164
- [Background] Grimble GK. Adverse gastrointestinal effects of arginine and related amino acids. J Nutr. 2007 Jun;137(6 Suppl 2):1693S-1701S. doi: 10.1093/jn/137.6.1693S. PMID 17513449
- [Background] Moinard C, Nicolis I, Neveux N, Darquy S, Benazeth S, Cynober L. Dose-ranging effects of citrulline administration on plasma amino acids and hormonal patterns in healthy subjects: the Citrudose pharmacokinetic study. Br J Nutr. 2008 Apr;99(4):855-62. doi: 10.1017/S0007114507841110. Epub 2007 Oct 22. PMID 17953788
- [Background] Papadia C, Sherwood RA, Kalantzis C, Wallis K, Volta U, Fiorini E, Forbes A. Plasma citrulline concentration: a reliable marker of small bowel absorptive capacity independent of intestinal inflammation. Am J Gastroenterol. 2007 Jul;102(7):1474-82. doi: 10.1111/j.1572-0241.2007.01239.x. Epub 2007 Apr 24. PMID 17459021
- [Background] Sureda A, Cordova A, Ferrer MD, Tauler P, Perez G, Tur JA, Pons A. Effects of L-citrulline oral supplementation on polymorphonuclear neutrophils oxidative burst and nitric oxide production after exercise. Free Radic Res. 2009 Sep;43(9):828-35. doi: 10.1080/10715760903071664. Epub 2009 Jul 6. PMID 19585317
- [Background] Bailey SJ, Blackwell JR, Lord T, Vanhatalo A, Winyard PG, Jones AM. l-Citrulline supplementation improves O2 uptake kinetics and high-intensity exercise performance in humans. J Appl Physiol (1985). 2015 Aug 15;119(4):385-95. doi: 10.1152/japplphysiol.00192.2014. Epub 2015 May 28. PMID 26023227
- [Background] Keteyian SJ. Exercise training in congestive heart failure: risks and benefits. Prog Cardiovasc Dis. 2011 May-Jun;53(6):419-28. doi: 10.1016/j.pcad.2011.02.005. PMID 21545928
- [Background] Acanfora D, Scicchitano P, Casucci G, Lanzillo B, Capuano N, Furgi G, Acanfora C, Longobardi M, Incalzi RA, Piscosquito G, Ciccone MM. Exercise training effects on elderly and middle-age patients with chronic heart failure after acute decompensation: A randomized, controlled trial. Int J Cardiol. 2016 Dec 15;225:313-323. doi: 10.1016/j.ijcard.2016.10.026. Epub 2016 Oct 11. PMID 27750131
- [Background] O'Connor CM, Whellan DJ, Lee KL, Keteyian SJ, Cooper LS, Ellis SJ, Leifer ES, Kraus WE, Kitzman DW, Blumenthal JA, Rendall DS, Miller NH, Fleg JL, Schulman KA, McKelvie RS, Zannad F, Pina IL; HF-ACTION Investigators. Efficacy and safety of exercise training in patients with chronic heart failure: HF-ACTION randomized controlled trial. JAMA. 2009 Apr 8;301(14):1439-50. doi: 10.1001/jama.2009.454. PMID 19351941
- [Background] Laratta CR, van Eeden S. Acute exacerbation of chronic obstructive pulmonary disease: cardiovascular links. Biomed Res Int. 2014;2014:528789. doi: 10.1155/2014/528789. Epub 2014 Mar 2. PMID 24724085